CLINICAL TRIAL: NCT02719262
Title: Workplace Intervention and Reduced Ambient Melamine Exposure and Renal Damage in Melamine Tableware Manufacturing Workers
Brief Title: Reduced of Ambient Melamine Exposure by Melamine Workplace Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Tsang Wu, Director of Center of Environmental & Occupational Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMU-F105002
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Environmental Exposure
Keywords: Melamine; Renal damage; Workplace intervention

STUDY DESIGN:
Intervention Model Description: Install local ventilation or not
Masking Description: Blinded by lab. persons who analyzed biomarkers
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): installing ventilation in the workplace
  Interventions: Device: installing ventilation in the workplace

INTERVENTIONS:
Device: installing ventilation in the workplace — Environmental improvement by installing/ exhaust ventilation (FUDIN SYSTEM ENGINEERING CO.,LTD.)

SUMMARY:
The investigators recent study has found that ambient melamine exposure can cause the increase of biomarkers of renal tubular injury in melamine manufacturing workers. Thus, in this year, the investigators will examine whether the intervention by installing ventilation in the workplace and providing personal protective equipment and education can decrease ambient melamine exposure and further decrease urinary biomarkers of renal tubular injury such as N-acetyl β-D-glucosaminidase (NAG) and β2-microglobulin (β2-MG).

DETAILED DESCRIPTION:
The investigators through intervention trial design to examine whether the use of ventilation in the workplace can decrease ambient melamine exposure, oxidative stress markers (such as 8-hydoxy-2-deoxyguanosine, malondialdehyde)and indicators of early renal damage (such as N-acetyl β-D-glucosaminidase, microalbumin and β2-microglobulin). The one week before intervention and the second week after intervention, the volunteers were asked to collect their urine samples for one consecutive week during mornings and afternoons. Blood samples were taken on Fridays morning, workplace air was sampled for 5 consecutive days. Then the investigators continued to trace the melamine concentration change of volunteers and workplace every three-month intervals after intervention, and blood samples were taken on 12th and 24th month.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult over age of 20 years

Exclusion Criteria:

* any hormone treatment or major chronic diseases (such as: cancer, hypertension, diabetes, chronic kidney disease and chronic liver disease) and patients with urinary calculi or family history of urinary calculi

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Change of melamine in air and in urine | 1 weeks
  Measured by liquid chromatograph/tandem mass spectrometry

SECONDARY OUTCOMES:
Oxidative stress markers 8-hydoxy-2-deoxyguanosine (8-OHdG) | 6 months
  Urinary 8-OHdG concentration was measured using a validated method of online SPE LC-MS/MS.
oxidative stress markers malondialdehyde (MDA) | 6 months
  Urinary MDA was measured by using HPLC-FL with a reversed-phase column.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsang Wu, MD, ScD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided